CLINICAL TRIAL: NCT04874233
Title: A 61-day Randomized, Double Blind, Placebo-controlled Trial to Assess the Safety and Efficacy of Three Doses of HU6 in Subjects With Elevated Liver Fat and High Body Mass Index (28 to 45 kg/m2)
Brief Title: Phase 2a Study of HU6 in Subjects With Elevated Liver Fat and High BMI Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rivus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIV-HU6-203
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-04

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Treatment: HU6 150 mg; N = 20 (Active Comparator): HU6 is Active Study Drug
  Interventions: Drug: HU6
- Active Treatment: HU6 300 mg; N = 20 (Active Comparator): HU6 is Active Study Drug
  Interventions: Drug: HU6
- Active Treatment: HU6 450 mg; N = 20 (Active Comparator): HU6 is Active Study Drug
  Interventions: Drug: HU6
- Placebo Comparator Non-active study drug N = 20 (Placebo Comparator): Non-active Study Drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HU6 — HU6 is active study drug
  Arms: Active Treatment: HU6 150 mg; N = 20; Active Treatment: HU6 300 mg; N = 20; Active Treatment: HU6 450 mg; N = 20
Drug: Placebo — Non-active study drug N = 20
  Arms: Placebo Comparator Non-active study drug N = 20

SUMMARY:
This is a Phase 2a, randomized, parallel-group, placebo-controlled, double-blind, repeated-dose study to evaluate the safety and efficacy of three oral dose levels of HU6 compared to placebo over the course of 61 days in subjects with high BMI and evidence of elevated liver fat.

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, parallel-group, placebo-controlled, double-blind, repeated-dose study to evaluate the safety and efficacy of three oral dose levels of HU6 compared to placebo over the course of 61 days in subjects with high BMI and evidence of elevated liver fat.

Subjects will be screened over a 45 day period to determine their eligibility based on specific history, physical, laboratory and imaging evaluations as per the Schedule of Assessments. Due to scheduling of the procedures, multiple visits will likely be necessary to complete the screening process. However, if all screening assessments and procedures, including the MRI, can be completed within 30 days of the first dose, then a single screening visit is permissible.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult male or females, 28 to 65 years of age (inclusive) at the time of informed consent with BMI between 28.0 and 45.0 kg/m2 (inclusive).

  1. Female subjects of childbearing potential must be non-lactating, not pregnant as confirmed by a negative urine pregnancy test at Screening and agree to continue using an effective method of contraception for at least 4 weeks or barrier method for 2 weeks prior to first study drug administration until 30 days after the last dose of study drug (Section 8.3.2).
  2. Female subjects of childbearing potential must not donate ova during the study and for at least 30 days after the last dose of study drug.
  3. Female subjects of non-childbearing potential must be surgically sterile (e.g., hysterectomy, bilateral tubal ligation, oophorectomy) or postmenopausal (no menses for >1 year with follicle stimulating hormone (FSH) >40 U/L at Screening).
  4. Male subjects who have not had a vasectomy and/or subjects who have had a vasectomy but have not had 2 post surgery negative tests for sperm must agree to use an acceptable method of contraception from time of first dose of study drug until 30 days after the last dose of the study drug, and to not donate sperm during the study and for at least 30 days after the last dose of study drug.

     2. Inclusion as per investigator assessment of general medical status and as documented by medical history, physical examination, vital sign assessments, 12-lead ECG, clinical laboratory assessments, and general observations.

  <!-- -->

  1. Subjects must be on stable doses of medications for underlying obesity-related conditions for at least 2 months prior to screening.
  2. Subjects with diabetes may be treated with metformin, DPP-4 inhibitors, or sulfonylureas, but must be on stable doses for at least 2 months prior to screening.
  3. At Screening, certain laboratory values may be outside the reference range if commensurate with the underlying obesity or associated metabolic dysfunction in the eligible subject (for example, dyslipidemia and hyperglycemia), unless these abnormalities suggest an underlying condition which may impact subject safety in the trial or interfere with the evaluation of HU6 or affect interpretation of the study results.
  4. Abnormalities or deviations outside the normal ranges for other assessments that are considered clinically significant by the Investigator (clinical laboratory tests, ECG, vital signs, physical examination) may be repeated once at the discretion of the Investigator(s). Results that continue to be outside the normal ranges must be judged by the investigator to be not clinically significant and acceptable for study participation.
  5. Subjects with elevation of unconjugated bilirubin due to presumptive Gilbert's syndrome are permissible.
  6. Subject must be euthyroid as assessed by a thyroid profile utilizing thyroid stimulating hormone (TSH) and free thyroxine (T4) testing at screening. Subjects with a stable history of thyroid disease and who have been on stable doses of thyroid medications for a minimum of 4 months can be enrolled.

     3. Fibroscan® CAP score>300 dB/m. 4. ≥8% liver fat by MRI-PDFF. 5. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

     6. Willing and able to comply with the requirements of the study protocol.

     Exclusion Criteria:

Subjects will be excluded from the study if any of the following criteria are met:

1. Insulin-controlled diabetes.
2. Pregnant or breastfeeding or plans to become pregnant.
3. Intolerance to Magnetic Resonance Imaging (MRI) or with conditions contraindicated for MRI procedures including but not limited to inability to fit into MRI scanner or surgical clips/metallic implants/shrapnel. Subjects must not be claustrophobic, have a history of claustrophobia, or intolerance of closed or small spaces.
4. Weight gain or loss >5% in 3 months prior to study or >10% in 6 months prior to screening.
5. History of lap banding, intragastric balloon, duodenal-jejunal sleeve, or bariatric surgery within 5 years of screening, plans for bariatric surgery prior to conclusion of study participation, or plans to lose weight during this study either through a special diet, exercise program or both.
6. History of malignant hyperthermia.
7. History of chronic serious recurrent skin rashes of unknown cause.
8. History of or current clinically significant cardiovascular disease including but not limited to transient ischemic attack, stroke, cardiac arrhythmias, syncope, unstable angina, myocardial infarction in the 6 months prior to screening, congestive heart failure, or uncontrolled hypertension. (Uncontrolled hypertension is defined as a systolic blood pressure ≥160 mmHg or a diastolic blood pressure ≥100 mmHg based on an average of three resting determinations in the sitting position with an appropriately sized cuff).
9. Resting heart rate <45 or >110 bpm.
10. On screening ECG or by history:

    1. A marked baseline prolongation of QT/QTcF interval (e.g., repeated demonstration of a QTcF interval > 450 msec for males and >470 msec for females).
    2. A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or a family history of sudden cardiac death of unknown origin.
11. Kidney disease, kidney transplant, or estimated glomerular filtration rate (eGFR) <50 mL/min/1.73 m2 based on the CKD-EPI Creatinine Equation (NKF 2009; https://www.kidney.org/content/ckd-epi-creatinine-equation-2009).
12. Significant lung disease requiring chronic daily medication including chronic obstructive pulmonary disease (COPD), emphysema, pulmonary fibrosis, or asthma.
13. Untreated obesity hypoventilation syndrome (OHS) or obstructive sleep apnea (OSA).
14. History of or active (acute or chronic) liver disease other than nonalcoholic fatty liver disease (NAFLD)/ nonalcoholic steatohepatitis (NASH), such as but not limited to autoimmune liver disease, viral hepatitis, genetic hemochromatosis, primary biliary cirrhosis, Wilson disease, alpha-1-antitrypsin deficiency, alcohol liver disease, acute fatty liver of pregnancy or drug induced (including acetaminophen) liver disease.
15. History of or treatment for clinically significant gastroparesis, inflammatory bowel disease, or any surgery of the upper gastrointestinal tract with the exception of cholecystectomy, or minor gastric procedures that are approved by the medical monitor.
16. History of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy, or variceal bleeding.
17. History of acute pancreatitis within one year of screening or chronic pancreatitis of any cause.
18. Serum triglyceride concentrations exceeding 500 mg/dL.
19. HbA1c >9.0%.
20. Familial (mother/father/sibling) and/or personal history of retinal detachment any time in the past.
21. Any history of or current diagnosis of Glaucoma.
22. Evidence of the following on screening ophthalmologic examination:

    1. Peripheral retinal pathology requiring treatment, retinal tears, or lattice that require treatment.
    2. Diabetic retinopathy with macula exudates or macula edema as shown by optical coherence tomography (OCT) and examination.
    3. Any active macular disease that affects the vision, including macula pucker (epiretinal membrane) and macular degeneration.
    4. Visually significant cataract as determined by ophthalmologist.
    5. Any previous intravitreal injection of anti-VEGF agents for macular degeneration.
    6. History of prior vitrectomy.
23. History of malignant neoplasms within 5 years of screening, except for basal cell or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer that is not currently or expected to require radiation therapy, chemotherapy and/or surgical interventions or to initiate hormonal treatment.
24. History of organ transplantation.
25. Received a COVID-19 vaccine less than 1 week prior to dosing (Visit 2 / Day 1) and/or plans to receive a COVID-19 vaccine during the study period.
26. History of significant drug abuse within one year prior to Screening or frequent use of soft drugs (such as marijuana) within 3 months prior to the Screening visit, or hard drugs (such as cocaine, phencyclidine [PCP], opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
27. History of alcoholism in the last 2 years or current evidence of excessive alcohol consumption as assessed by screening evaluation using the Alcohol Use Disorders Identification Test (AUDIT, Thompson 2018 [Appendix A]), and history of regular alcohol consumption exceeding approximately 14 drinks/week for men and 7 drinks/week for women [1 drink = 4 ounces (120 mL) of wine or 12 ounces (360 mL) of beer or 1 ounce (30 mL) of hard liquor] within 6 months of Screening, as determined by the Investigator.
28. Positive urine drug screen for drugs of abuse or positive phosphatidylethanol (PEth) blood test result >25 ng/mL at Screening.
29. Current regular vaping or more than 5 cigarettes or the equivalent per week. Use of nicotine patches for smoking cessation is permitted.
30. Positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV1/2) antibody.
31. Neutropenia, defined as absolute neutrophil count ≤1000/μL.
32. Serum AST or ALT >5 x upper limit of normal (ULN) at screening. (One repeat test may be allowed within 7 days at the discretion of the Investigator).
33. Total bilirubin > ULN, unless due to Gilbert's syndrome or if considered normal variability in the absence of other clinically relevant liver impairment as approved by Medical Monitor.
34. International normalized ratio (INR) ≥1.3 at screening if there is other evidence of potential significant liver impairment.
35. Participation in another clinical trial at the time of screening or exposure to any investigational agent, including topical, within 30 days of screening or 5 half-lives, if half-life known.
36. No tattoo or body piercings during the course of the study. Any underlying physical or psychological medical condition that, in the opinion of the Investigator or sponsor, would make it unlikely that the subject is able comply with the study requirements or would be unable to complete the study.
37. Any condition that the investigator believes would interfere with his/her ability to provide written informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.
38. Known or potential hypersensitivity to HU6 or its excipients.

    Prohibited Medications (Current Use):
39. Any herbal supplement, over the counter drug, mail order or prescription drug for weight loss.
40. Prescription or over the counter stimulants including: dextroamphetamine/Dexedrine, dextroamphetamine/amphetamine combination product/Adderall, or methylphenidate (Ritalin®, Concerta®).
41. Thiazolidinediones (TZD): pioglitazone/Actos, rosiglitazone/Avandia.
42. Glucagon-like peptide 1 (GLP1) agonists: exenatide/Byetta/Bydureon, lixisenatide/Adlyxin, liraglutide/Victoza, dulaglutide/Trulicity, semaglutide/Ozempic.
43. Sodium-glucose cotransporter-2 (SGLT2) inhibitors: canagliflozin/Invokana, dapagliflozin/Farxiga, empagliflozin/Jardiance, ertugliflozin/Steglatro.
44. Vitamin E: use of ursodiol or high dose vitamin E >400 IU/day for at least one month within in the last 6 months or started high dose vitamin E within last 3 months of screening.
45. Recent (within 3 months of screening) or current use of obeticholic acid/Ocaliva, systemic corticosteroids, methotrexate, tamoxifen, amiodarone, or long-term use of tetracyclines.
46. Warfarin, heparin, factor Xa inhibitors (dabigatran betrixaban edoxaban, apixaban, and rivaroxaban).
47. Concomitant medications that prolong the QT/QTc interval and are known to be associated with increased risk of Torsade des pointes as identified in the https://crediblemeds.org/ website list category of 'Known Risk' (Appendix B).
48. Products with cannabidiol (CBD).

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Eastenson, Principal Investigator — Prism Clinic Research
Locations (1):
- Prism Clinical Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureddin M, Khan S, Portell F, Jorkasky D, Dennis J, Khan O, Johansson L, Johansson E, Sanyal AJ. Safety and efficacy of once-daily HU6 versus placebo in people with non-alcoholic fatty liver disease and high BMI: a randomised, double-blind, placebo-controlled, phase 2a trial. Lancet Gastroenterol Hepatol. 2023 Dec;8(12):1094-1105. doi: 10.1016/S2468-1253(23)00198-X. Epub 2023 Oct 5. PMID 37806314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Start: April 19,2021, Completion: November 30,2021, Study Completion: December 15,2021 at one site
Groups:
- Active Treatment: HU6 150 mg: Active Treatment: HU6 150 mg; HU6 is active study drug
- Active Treatment: HU6 300 mg: Active Treatment: HU6 300 mg; HU6 is active study drug
- Active Treatment: HU6 450 mg: Active Treatment: HU6 450 mg; HU6 is active study drug
- Placebo Comparator Non-active Study Drug: Placebo Comparator Non-active study drug Placebo: Non-active study drug
Period: Overall Study
Arm/Group | Active Treatment: HU6 150 mg | Active Treatment: HU6 300 mg | Active Treatment: HU6 450 mg | Placebo Comparator Non-active Study Drug
Started | 20 | 21 | 19 | 20
Completed | 18 | 20 | 19 | 17
Not Completed | 2 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Active: HU6 150mg: HU6 150mg is active Study Drug
- Active: HU6 300mg: HU6 300mg is active study drug
- Active: HU6 450mg: HU6 450 mg is active study drug
- Placebo Comparator: Non-active study drug
- Total: Total of all reporting groups
Arm/Group | Active: HU6 150mg | Active: HU6 300mg | Active: HU6 450mg | Placebo Comparator | Total
Number analyzed (Participants) | 20 | 21 | 19 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.31) | 47.1 (6.78) | 46.7 (10.04) | 50.7 (9.24) | 47.7 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 8 | 9 | 39
  Male | 10 | 9 | 11 | 11 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 0 | 0 | 4
  Not Hispanic or Latino | 19 | 18 | 19 | 20 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 4 | 0 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 15 | 19 | 17 | 17 | 68
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Liver fat content, as assessed by MRI-PDFF [Mean (Standard Deviation); unit: percentage of liver fat mass] | 18.6 (6.9) | 18.0 (8.2) | 17.3 (8.2) | 15.9 (5.9) | 17.7 (7.23)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change From Baseline in Liver Fat Content as Assessed by MRI-PDFF
Description: Percentage of Change from Baseline in Liver Fat Content as Assessed by MRI-PDFF at Day 61
Time Frame: Baseline and 61 days;
Population: For HU6 450mg, 19 participants were randomized, but 18 was the number of participants analyzed.
  Percent change from baseline=(Value at Day 61/Value at baseline x 100%)
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Active Treatment: HU6 300 mg;: Active Treatment: HU6 300 mg; HU6 is active study drug
- Active Treatment: HU6 450 mg;: Active Treatment: HU6 450 mg; HU6 is active study drug
- Placebo Comparator Non-active Study Drug: Placebo Comparator Non-active study drug; Placebo: Non-active study drug
Arm/Group | Active Treatment: HU6 150 mg | Active Treatment: HU6 300 mg; | Active Treatment: HU6 450 mg; | Placebo Comparator Non-active Study Drug
Number analyzed (Participants) | 20 | 21 | 18 | 20
percentage of change | -26.8 (17.4) | -35.6 (13.8) | -33.0 (18.4) | 5.4 (19.8)

ADVERSE EVENTS:
Time Frame: 61 days of dosing
Groups:
- Active: HU6 150mg; Active: HU6 300mg; Active: HU6 450mg: HU6 is active Study Drug
Arm/Group | Active: HU6 150mg | Active: HU6 300mg | Active: HU6 450mg | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 13/20 | 17/21 | 16/19 | 11/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active: HU6 150mg (N=20) | Active: HU6 300mg (N=21) | Active: HU6 450mg (N=19) | Placebo Comparator (N=20)
Flushing (Vascular disorders) | 3 | 8 | 8 | 2
Hot Flush (Vascular disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 6 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 2 | 2 | 3 | 1
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 3
Presyncope (Nervous system disorders) | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 1 | 2
Pyrexia (General disorders) | 0 | 2 | 1 | 2
Vessel puncture site haemorrhage (General disorders) | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 2 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04874233/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04874233/SAP_001.pdf